CLINICAL TRIAL: NCT05939661
Title: A Multicenter Single-arm Phase 2 Study to Evaluate Safety and Efficacy of the Total Neoadjuvant Therapy of Short Course Radiation Therapy Followed by Neoadjuvant Oxaliplatin/Fluorouracil-based Chemotherapy (CAPOX) for cT2 Rectal Cancer.
Brief Title: A Multicenter Single-arm P2 to Evaluate Safety and Efficacy of the Total Neoadjuvant Therapy for cT2 Rectal Cancer
Acronym: AMBITION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Osaka University (Other)
Responsible Party: Principal Investigator, Mamoru Uemura, Department of Gastroenterological Surgery, Osaka University Graduate School of Medicine, Osaka University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: jRCTs051230014
Record Dates: First submitted 2023-06-25; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Rectal Cancer
Keywords: total neoadjuvant therapy; neadjuvant chemotherapy; organ preservation; watch and wait; radiation; surgery; total mesorectum excision
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiation; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: RT→Chemo→Surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TNT (Experimental): Neoadjuvant radiation therapy : 5Gyx5 Neoadjuvant chemo therapy : CAPOX (Oxaliplatin 130mg/m2, Capecitabine2000mg/m2/day, d1-14, 3week)x6cycles Operation: Total methorectum excision wiht radical lymph node dissection
  Interventions: Radiation: Radiation; Drug: Chemotherapy; Procedure: Surgery

INTERVENTIONS:
Radiation: Radiation — Neoadjuvant radiation therapy : 5Gyx5
Drug: Chemotherapy — CAPOX (Oxaliplatin 130mg/m2, Capecitabine2000mg/m2/day, d1-14, 3week)x6cycles
Procedure: Surgery — Operation: Total methorectum excision wiht radical lymph node dissection

SUMMARY:
A multicenter single-arm phase 2 study to evaluate safety and efficacy of the total neoadjuvant therapy of short course radiation therapy followed by neoadjuvant oxaliplatin/fluorouracil-based chemotherapy (CAPOX) for cT2 rectal cancer

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of preoperative radiation therapy followed by preoperative chemotherapy and surgery for T2 advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient has been fully informed of the contents of the study and has given written consent.

  2. The patient has adenocarcinoma of the rectum confirmed by histological examination.

  3. No distant metastases are detected on imaging studies, and radical resection is clinically feasible.

  4. Age of 20 years or older on the date of consent. 5. ECOG Performance Status (PS) is 0 - 1 (PS 0 for age 71 years or older on the date of consent).

  6. Previously untreated rectal cancer with the lower margin of the tumor within 12 cm of the anal verge (AV).

  7. Patients with cT2N0M0 in the diagnosis before starting treatment (a lymph node with a short diameter of 7 mm or more is considered positive).

The conditions for lymph node metastasis shall be as follows. Contrast-enhanced CT or MRI (plain or contrast-enhanced) with a slice width of 5 mm or less.

(i) Short diameter of 10 mm or more (ii) Short diameter of 7 mm or more and one or more of the following a) to c) are met

(a) Edge irregularity (b) Low signal area with internal heterogeneity on MRI (c) Circular (long/short diameter ratio < 1.5) If contrast-enhanced CT is not possible due to contrast medium allergy, renal dysfunction, or bronchial asthma, simple CT is acceptable.

8. The following criteria for major organ function within 14 days prior to registration are met.

If more than one test result exists within this period, the most recent one should be used. No blood transfusions or hematopoietic factor products should be administered within 14 days prior to the test date.

1. Neutrophil count: greater than or equal to 1,500/mm3
2. Platelet count: >= 10.0 x 104 /mm3
3. Hemoglobin concentration: >=9.0 g/dL
4. Total bilirubin: 1.5 times or less than the upper limit of the institutional standard
5. AST, ALT, ALP: 2.5 times or less than the upper limit of the institutional standard
6. Serum creatinine: 1.5 times or less than the upper limit of the institutional standard or creatinine clearance: 45 mL/min or more

Exclusion Criteria:

* 1. underwent treatment by any of the following within a certain period of time prior to initiation of protocol therapy

  1. extensive surgery (excluding CV port placement) within 4 weeks
  2. Any anticancer therapy within 4 weeks
  3. Radiation within 4 weeks 2. concomitant or pre-existing severe pulmonary disease (interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc.) 3. patients who have had a colonic stent implanted 4. patients with serious comorbidities (heart failure, renal failure, liver failure, bleeding peptic ulcer, intestinal paralysis, bowel obstruction, poorly controlled diabetes, etc.) 5. patients with active multiple overlapping cancers (synchronous multiple overlapping cancers or iatrogenic multiple overlapping cancers with a disease-free period of 5 years or less). However, carcinoma in situ (intraepithelial carcinoma) or intramucosal carcinoma that is considered curable by local treatment is not considered active multiple overlapping carcinoma.

     6. pregnant or lactating women, positive pregnancy test or unwillingness to use contraception 7. HBs antigen positive or HCV antibody positive. 8. has known human immunodeficiency virus (HIV) infection. 9. otherwise judged by the principal investigator or subinvestigator to be unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | through study completion, an average of 6 months
  pCR is evaluated by using the grading scale according to the Japanese Classification of Colorectal, Appendiceal, and Anal Carcinoma

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Osaka General Medical Center, Osaka
  - Osaka University Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No